CLINICAL TRIAL: NCT01488149
Title: Intrapartum Epidural Fentanyl and Breast-feeding in the Immediate Postpartum Period: a Prospective Cohort Study
Status: Withdrawn | Type: Observational
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: epidural fentanyl
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Maternal Anaesthesia and Analgesia Affecting Fetus or Newborn; Breast Feeding; Fentanyl; Bupivacaine; Nalbuphine
Keywords: Fentanyl; Bupivacaine; Nalbuphine
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recipients of intrapartum epidural analgesia
- Non-recipients of intrapartum epidural analgesia

SUMMARY:
Intrapartum epidural analgesia has been associated with adverse breastfeeding outcomes. One potential mechanism involves transfer of epidural fentanyl across the placenta and neonatal blood-brain barrier, where it can subsequently attenuate neonatal exhibition of feeding behaviors, such as latching and swallowing, during the immediate postpartum period. Vigorous feeding behavior during the first days of life is a significant predictor of long-term breastfeeding success at 3 and 6 months. In a randomized, controlled, double-blinded study, neonatal Neurologic and Adaptive Capacity Scores (NACS) were significantly lower when mothers received >150 mcg epidural fentanyl versus bupivacaine-only analgesia, and mean umbilical cord fentanyl concentration was significantly higher in the >150 mcg versus <150 mcg group.

The investigators hypothesize that epidural fentanyl-bupivacaine analgesia is significantly associated with decreased breastfeeding rates at hospital discharge and with neonatal deficits in latching onto the breast and swallowing during the first three hours of life, and that a significant dose-response relationship exists with respect to total micrograms fentanyl infused.

The investigators will perform a prospective cohort study of all parturients age 18+ at UHCMC over a three-month period, excluding those with multiples gestation, Cesarean section, or neonatal intensive care unit admission. From patient charts, the investigators will record the following variables: number of neonates delivered; type of delivery (spontaneous vaginal / operative vaginal / Cesarean section); whether the neonate was admitted to the intensive care unit; the mother's age, height, weight, gravity, parity, intention to breast-feed at the time of hospital admission, number of children previously breast-fed, and ethnicity; gestational age at the time of delivery; administration of oxytocin for labor augmentation and in what quantity; duration of active labor; antibiotic administration; neonatal APGAR scores at 1 and 5 minutes postpartum; and whether opioids or antibiotics were administered before and/or after the delivery and at what exact time. We will also record whether each patient received an epidural during labor and, if so, the duration of this epidural infusion and the total micrograms fentanyl delivered; neonatal feeding behavior as quantified by the LATCH scores assigned to each breast-feeding interaction that occurs on the postpartum care floor; whether the mother is breast-feeding her baby at the time of discharge from the hospital, and if not, then her primary reason for not doing so (as communicated during the standard postpartum lactation consultation); and how long mother and baby stayed in the hospital post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over

Exclusion Criteria:

* multiples gestation
* Cesarean section
* neonatal intensive care unit admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturients who deliver a single live neonate at UHCMC between February 2012 and June 2012
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Neonatal deficiency in latching on to the breast and/or audibly swallowing during feeding | First 5 hours postpartum
  Measured by the standardized LATCH scoring system

SECONDARY OUTCOMES:
Likelihood of breast-feeding at the time of hospital discharge, either exclusively or with bottle supplementation | Time of discharge from hospital (on average, 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L Szabo, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Baumgarder DJ, Muehl P, Fischer M, Pribbenow B. Effect of labor epidural anesthesia on breast-feeding of healthy full-term newborns delivered vaginally. J Am Board Fam Pract. 2003 Jan-Feb;16(1):7-13. doi: 10.3122/jabfm.16.1.7. PMID 12583645
- [Background] Beilin Y, Bodian CA, Weiser J, Hossain S, Arnold I, Feierman DE, Martin G, Holzman I. Effect of labor epidural analgesia with and without fentanyl on infant breast-feeding: a prospective, randomized, double-blind study. Anesthesiology. 2005 Dec;103(6):1211-7. doi: 10.1097/00000542-200512000-00016. PMID 16306734
- [Background] Henderson JJ, Dickinson JE, Evans SF, McDonald SJ, Paech MJ. Impact of intrapartum epidural analgesia on breast-feeding duration. Aust N Z J Obstet Gynaecol. 2003 Oct;43(5):372-7. doi: 10.1046/j.0004-8666.2003.t01-1-00117.x. PMID 14717315
- [Background] Wiklund I, Norman M, Uvnas-Moberg K, Ransjo-Arvidson AB, Andolf E. Epidural analgesia: breast-feeding success and related factors. Midwifery. 2009 Apr;25(2):e31-8. doi: 10.1016/j.midw.2007.07.005. Epub 2007 Nov 5. PMID 17980469
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525